CLINICAL TRIAL: NCT03635918
Title: Extensive Prospective Validation Study of the NightOwl Home Sleep Apnea Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ectosense NV (Industry)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17/034-11/06/2018
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NightOwl HSAT (Other): Patient undergoes a NightOwl sleep apnea test whilst simultaneously undergoing a sleep study with a Type I sleep monitor (Lab-PSG) and optionally a benchmark HSAT monitor.
  Interventions: Device: NightOwl HSAT

INTERVENTIONS:
Device: NightOwl HSAT — Patient wears the NightOwl sensor device

SUMMARY:
Extensive Prospective validation study of the NightOwl, a Type IV home sleep apnea test (HSAT), compared to traditional PSG and HSAT monitors.

DETAILED DESCRIPTION:
The purpose of this prospective validation study is the evaluation of the accuracy of the NightOwl HSAT to derive parameters relevant for the diagnosis of sleep apnea. The NightOwl HSAT comprises a finger or forehead mounted sensor and an automated analytics software. The sensor measures double-wavelength photo-plethysmography and accelerometry. The analytics software automatically interprets the sensor data and derives a measure of sympathetic activation of the autonomic nervous system, oxygen saturation, instantaneous pulse rate and activity. For each patient in the cohort, the AHI derived by the NightOwl will be compared to that of the Type I sleep monitor (in-lab PSG), which will acquire data simultaneously during the diagnostic night of the patient referred to the sleep lab for a polysomnography. On a randomly selected subset of patients, a benchmark HSAT will additionally be applied for comparison of its automated AHI derivation to that of the NightOwl.

ELIGIBILITY:
Inclusion Criteria:

* indication for a sleep study

Exclusion Criteria:

* Mentally disabled people

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-09-15 (Estimated); Study Completion 2019-09-15 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | For each included patient, the outcome measure will be assessed immediately after analysis of that patient's data by the NightOwl HSAT software
  Comparison of the AHI derived from the NightOwl HSAT to that of the benchmark PSG and HSAT monitors.

SECONDARY OUTCOMES:
Sleep-wake discrimination | For each included patient, the outcome measure will be assessed immediately after analysis of that patient's data by the NightOwl HSAT software
  Comparison of the sleep-wake discrimination derived from the NightOwl HSAT to that of the benchmark PSG and HSAT monitors.

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Massie, ir., Study Director — Ectosense NV
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No